CLINICAL TRIAL: NCT02272920
Title: Combined Treatment With Percutaneous Coronary Intervention and Renal Denervation in Hypertensive Patients With Acute Coronary Syndromes.
Brief Title: PCI and Renal Denervation in Hypertensive Patients With Acute Coronary Syndromes
Acronym: COMBI-RDN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Elmir Omerovic, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 538-13
Record Dates: First submitted 2014-09-11; First posted 2014-10-23 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Acute Myocardial Infarction
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation (Experimental): One procedure will be performed using one of the CE-marked devices for renal denervation: Medtronic Symplicity Flex, Medtronic Symplicity Spyral or St Jude EnligHTN.
  Renal denervation is performed within seven days after PCI in patients with acute myocardial infarction and hypertension.
  Interventions: Procedure: Renal denervation
- Control: Standard of care (No Intervention): Standard-of-care follow-up after ACS. Including nurse and physician out-patient visits.

INTERVENTIONS:
Procedure: Renal denervation — Medtronic Symplicity Flex, Medtronic Symplicity Spyral, or St Jude EnligHTN.
  Arms: Renal denervation

SUMMARY:
Research hypothesis:

Is the treatment with renal denervation (RDN) early post ACS safe and effective and does it leads to improved cardiac function and attenuation of pathologic left ventricular remodelling? In a following study, the hypothesis will be tested in a larger ACS population with major adverse cardiovascular events (MACE) after ACS as the endpoint.

Rationale for conducting this study:

ACS i.e. ST-elevation myocardial infarction (STEMI) and non- ST-elevation myocardial infarction (non-STEMI) are the most important causes of morbidity and mortality in western societies. Hypertension is a major risk factor for development of ACS and heart failure but it also worsens the prognosis in patients after ACS. Our research highlights the combination therapy of PCI and RDN in an ACS patient population with simultaneous hypertension.

Primary objective:

The primary objective of this study is to establish safety and efficacy of combined treatment with PCI and renal denervation (RDN) in hypertensive patients with acute coronary syndromes (STEMI and non-STEMI ) having ventricular mass after 4 months as the primary variable.

Endpoints:

The primary end point is change in left ventricular mass (LVM) at 4 months evaluated by magnetic resonance imaging (MRI).

Secondary endpoints:, blood pressure (office and 24-h ABPM), and left ventricular volumes and ejection fraction.

DETAILED DESCRIPTION:
The sympathetic nervous system plays a crucial role in the development and progression of hypertension and its adverse consequences. Despite the availability of numerous effective pharmacologic treatments, adequate blood pressure control is not achieved in a large number of subjects. Patients with essential hypertension generally have increased efferent sympathetic drive to the kidneys and an increased rate of sympathetic-nerve firing, possibly modulated by afferent signalling from renal sensory nerves. Recently developed endovascular catheter technology enables selective denervation of the human kidney. A safety and feasibility trial of this procedure identified substantial reductions of blood pressure without substantial procedure-related complications. The therapeutic value seems to be present not only in hypertension but may also be of interest in many clinical conditions e.g. heart failure, chronic end-stage renal disease and insulin resistance and diabetes.

The present study (COMBI-RDN) is a randomised clinical trial in 40 patients to investigate safety and efficacy of the combination of Percutan Coronar Interventiom (PCI) and renal denervation (RDN) where RDN is performed early after acute coronary syndrome (ACS). This study is considered a pilot study to evaluate efficacy and safety in patients with ACS. In a second phase there will be a randomised, multicenter study in approximately 2500 patients to demonstrate whether RDN early post ACS could decrease major adverse cardiovascular events in hypertensive patients with ACS.

Research hypothesis Is the treatment with renal denervation (RDN) early post ACS safe and effective and does it leads to improved cardiac function and attenuation of pathologic left ventricular remodelling?

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male aged 18-80 years
3. Patients with ACS, i.e. STEMI, non-STEMI, treated with PCI
4. Medical history of treated (ongoing) hypertension, or hypertension discovered at the time of ACS, and office SBP >140 despite treatment with three antihypertensive drugs.
5. Ejection fraction >40%.

Exclusion Criteria:

1. Increased risk of pathological bleedings
2. Office systolic blood pressure <120
3. Renal artery abnormalities.
4. eGFR <30 mL/min
5. ICD or pacemaker, or any other metallic implant not compatible with MRI
6. Estimated survival time <1 year
7. Not oriented to person, place and time
8. Inability to understand given information about the study
9. Fertile female

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Left ventricular remodelling | At 4 months.
  Change in left ventricular mass and volumes, as measured by magnetic resonance. Comparing intervention and control group.

SECONDARY OUTCOMES:
Office and 24-h ambulatory blood pressure | At 4 months after renal denervation.
  Change in blood pressure. Comparing intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Bert Andersson, Prof MD, Principal Investigator — Dept of Cardiology, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden